CLINICAL TRIAL: NCT01790126
Title: The Role of Highly Selective Androgen Receptor (AR) Targeted Therapy in Men With Biochemically Relapsed Hormone Sensitive Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR103305; ARN-509-002
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer
Keywords: Men with Biochemically Relapsed Hormone Sensitive Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Gonadotropin-Releasing Hormone; luprolide acetate gel depot; Leuprolide; Goserelin; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- ARN-509 (Active Comparator): ARN-509 Tablets, 240 mg/day administered orally
  Interventions: Drug: ARN-509
- LHRH agonist + ARN-509 (Active Comparator): Choice of LHRHa per investigator discretion/site practice guidelines (e.g, Eligard®, Zoladex®, Lupron Depot®, Trelstar®) and ARN-509 Tablets, 240 mg/day administered orally
  Interventions: Drug: ARN-509; Drug: LHRH Agonist
- LHRH agonist (Active Comparator): Choice of LHRHa per investigator discretion/site practice guidelines (e.g., Eligard®, Zoladex®, Lupron Depot®, Trelstar®).
  Interventions: Drug: LHRH Agonist

INTERVENTIONS:
Drug: ARN-509
  Arms: ARN-509; LHRH agonist + ARN-509
Drug: LHRH Agonist
  Other Names: Eligard®; Lupron Depot®; Zoladex®; Trelstar®
  Arms: LHRH agonist; LHRH agonist + ARN-509

SUMMARY:
The proposed clinical trial will study the effects of 12 months of therapy with ARN-509 alone, or in combination with an LHRH agonist (LHRHa), each compared with LHRHa alone, in men with a rapidly rising serum PSA after prior definitive local therapy for prostate cancer. The endpoints selected reflect measurable short term effects of androgen deprivation therapy (ADT), including quality of life and several metabolic parameters. In addition, the relative effect of each treatment strategy on PSA suppression as well as testosterone recovery (and subsequent PSA progression) after 12 months of therapy will be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate
* Rising PSA after prior definitive local therapy (radical prostatectomy, external beam radiation, or brachytherapy) or combination of radical prostatectomy and radiotherapy with curative intent
* PSA doubling time less than or equal to 12 months
* No evidence of metastatic disease on imaging by whole body bone scan and computerized tomography (CT) or Magnetic Resonance Imaging (MRI) of the abdomen/pelvis within 6 weeks prior to randomization
* Minimum PSA 1.0 ng/mL if prior radical prostatectomy +/- adjuvant or salvage radiation; nadir + 2.0 ng/mL if prior RT without prior radical prostatectomy
* Prior androgen deprivation therapy (ADT) allowed if last dose was greater than (>) 6 months prior to randomization
* No prior androgen deprivation therapy (ADT) or anti-androgen for biochemical relapse
* Serum testosterone > 150 ng/dL at study entry
* No history of seizures or medical conditions which may lower seizure threshold

Key Exclusion Criteria:

* Use of 5-alpha reductase antagonist (i.e. finasteride, dutasteride) within 6 weeks prior to randomization
* Use of antiandrogen (e.g. flutamide, nilutamide, bicalutamide) within 6 weeks prior to randomization
* Prior bilateral orchiectomy
* Prior treatment with ADT for biochemically relapsed prostate cancer. Prior ADT as neo-adjuvant, concurrent, and/or adjuvant treatment following salvage radiation therapy or prostatectomy for biochemically relapsed disease is allowed provided last dose of ADT is greater than (>) 6 months prior to randomization and the Screening serum testosterone level is greater than or equal to (≥)150 ng/dL
* Use of systemic steroids at an equivalent dose of prednisone 5 mg/day or higher at randomization
* Any history of seizures or medical condition which lowers seizure threshold

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-03-04 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aragon Pharmaceuticals, Inc Clinical Trial, Study Director — Aragon Pharmaceuticals, Inc.
Locations (5):
- United States (5):
  - Scottsdale, Arizona
  - San Francisco, California
  - Chicago, Illinois
  - Portland, Oregon
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Luteinizing Hormone Releasing Hormone Agonist (LHRHa): Participants received LHRHa injections either subcutaneously or intramuscularly as per investigator discretion/site practice guidelines up to 12 months, or shorter duration if evidence of prostate-specific antigen (PSA)/radiographic progression or unacceptable toxicity during protocol therapy or participant/physician withdrawal from the study.
- Apalutamide: Participants received apalutamide, 240 milligram (mg) soft-gel capsules (8*30 mg capsules) per day orally up to 12 months, or shorter duration if evidence of PSA/radiographic progression or unacceptable toxicity during protocol therapy or participant/physician withdrawal from the study. With Amendment 7, participants who were receiving the apalutamide soft-gel capsules were switched to the apalutamide tablet formulation (4*60 mg tablets).
- LHRHa + Apalutamide: Participants received LHRHa injections either subcutaneously or intramuscularly as per investigator discretion/site practice guidelines and apalutamide 240 mg soft-gel capsules per day orally up to 12 months, or shorter duration if evidence of PSA/radiographic progression or unacceptable toxicity during protocol therapy or participant/physician withdrawal from the study. With Amendment 7, participants who were receiving the apalutamide soft-gel capsules were switched to the apalutamide tablet formulation (4*60 mg tablets).
Period: Overall Study
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Started | 30 | 29 | 31
Treated | 29 | 29 | 31
Completed | 0 | 0 | 0
Not Completed | 30 | 29 | 31
Not completed — PSA Progression | 12 | 16 | 16
Not completed — Other | 5 | 4 | 8
Not completed — Initiation of Non-Protocol Therapy | 3 | 4 | 2
Not completed — Withdrawal by Physician | 1 | 1 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Radiographic Progression | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide | Total
Number analyzed (Participants) | 30 | 29 | 31 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (6.51) | 66.1 (6.18) | 67.5 (6.67) | 67.0 (6.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 30 | 29 | 31 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 3
  Not Hispanic or Latino | 30 | 26 | 30 | 86
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 26 | 26 | 29 | 81
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 30 | 29 | 31 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy - Prostate (FACT-P) Total Score at 12 Months
Description: FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment. It is a combination of the FACT- General + the Prostate Cancer Subscale (PCS). The FACT-General (FACT-G) is a 27 item Quality of Life (QoL) measure that provides a total score as well as subscale scores: Physical (0-28), Functional (0-28), Social (0-28), and Emotional Well-being (0-24). The total score range is between 1-108, higher scores indicates better for total score and subscale scores. PCS is a 12-item prostate cancer subscale that asks about symptoms and problems specific to prostate cancer (Range 0-48, higher scores better). The FACT-P total score is the sum of all 5 subscale scores of the FACT-P questionnaire and ranges from 0-156. Higher scores indicate higher degree of functioning and better quality of life.
Time Frame: Baseline, at 12 months
Population: The intent-to-treat (ITT) population included all randomized participants and was classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 30 | 29 | 31
Units on a scale | -8.04 (2.40) | -6.60 (2.53) | -9.42 (2.30)

2. Secondary Outcome: Change From Baseline in FACT-P Total Score at 3 and 24 Months
Description: as for outcome 1
Time Frame: Baseline, at 3 and 24 months
Population: The ITT population included all randomized participants and was classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 30 | 29 | 31
Units on a scale
  Change at 3 months | -2.62 (2.49) | -4.80 (2.45) | -6.72 (2.29)
  Change at 24 months | -4.43 (2.91) | 1.84 (3.17) | -1.87 (2.59)

3. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Score at 3, 12 and 24 Months
Description: EORTC QLQ-C30 is a 30 items self-reporting questionnaire resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 Global Health Status (GHS) scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Questionnaire includes 28 items with 4-point Likert type responses from "1-not at all" to "4-very much" to assess functioning and symptoms; 2 items with 7-point Likert scales (1= poor and 7= excellent) for global health and overall health related quality of life. Scores are transformed to 0 to 100 scale, with higher scores representing better GHS, better functioning, and more symptoms.
Time Frame: Baseline, at 3, 12 and 24 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 30 | 29 | 31
Units on a scale
  Appetite loss: Change at 3 months | 2.80 (2.84) | 3.43 (2.75) | 8.04 (2.48)
  Appetite loss: Change at 12 months | 3.49 (3.34) | 4.87 (3.51) | 5.70 (3.09)
  Appetite loss: Change at 24 months | -2.29 (4.05) | -2.50 (4.35) | 5.28 (3.29)
  Cognitive functioning: Change at 3 months | -2.44 (3.69) | -6.83 (3.62) | -7.73 (3.28)
  Cognitive functioning: Change at 12 months | -2.21 (3.40) | -11.50 (3.58) | -8.27 (3.19)
  Cognitive functioning: Change at 24 months | -5.08 (4.16) | -12.71 (4.64) | -4.42 (3.55)
  Constipation: Change at 3 months | 2.90 (3.01) | -3.21 (2.94) | 3.45 (2.65)
  Constipation: Change at 12 months | 10.12 (3.18) | 0.27 (3.36) | 7.69 (2.96)
  Constipation: Change at 24 months | 0.45 (4.10) | 0.91 (4.43) | -0.10 (3.33)
  Diarrhoea: Change at 3 months | 5.99 (4.26) | 8.10 (4.20) | 8.09 (3.77)
  Diarrhoea: Change at 12 months | 0.02 (3.66) | 0.96 (3.87) | 3.28 (3.42)
  Diarrhoea: Change at 24 months | -0.35 (4.49) | -1.96 (4.97) | 4.38 (3.73)
  Dyspnoea: Change at 3 months | 6.42 (4.36) | 13.22 (4.29) | 12.85 (3.86)
  Dyspnoea: Change at 12 months | 4.45 (4.07) | 10.32 (4.34) | 9.49 (3.82)
  Dyspnoea: Change at 24 months | 11.16 (5.41) | 8.89 (5.86) | 7.34 (4.42)
  Emotional functioning: Change at 3 months | -0.81 (2.79) | -2.59 (2.73) | 1.41 (2.46)
  Emotional functioning: Change at 12 months | 1.39 (2.46) | 1.71 (2.60) | 3.84 (2.29)
  Emotional functioning: Change at 24 months | -0.60 (3.37) | 3.59 (3.67) | 3.13 (2.77)
  Fatigue: Change at 3 months | 11.40 (4.32) | 21.85 (4.30) | 22.40 (3.80)
  Fatigue: Change at 12 months | 15.29 (3.97) | 13.29 (4.22) | 19.80 (3.70)
  Fatigue: Change at 24 months | 11.33 (4.96) | 5.53 (5.49) | 5.81 (4.10)
  Financial difficulties: Change at 3 months | -5.91 (3.39) | -1.79 (3.33) | 2.49 (3.03)
  Financial difficulties: Change at 12 months | -6.26 (3.49) | 3.98 (3.70) | 3.90 (3.28)
  Financial difficulties: Change at 24 months | -10.69 (4.47) | -1.56 (4.88) | -3.90 (3.71)
  Global health status: Change at 3 months | -3.57 (3.45) | -10.30 (3.36) | -9.19 (3.01)
  Global health status: Change at 12 months | -4.90 (3.08) | -8.28 (3.23) | -6.08 (2.85)
  Global health status: Change at 24 months | -8.14 (4.14) | -3.73 (4.52) | -7.05 (3.39)
  Insomnia: Change at 3 months | 6.88 (6.18) | 5.31 (6.08) | 14.34 (5.46)
  Insomnia: Change at 12 months | 15.89 (5.46) | 2.71 (5.80) | 8.60 (5.12)
  Insomnia: Change at 24 months | 16.34 (6.96) | 2.49 (7.83) | -3.00 (5.76)
  Nausea and vomiting: Change at 3 months | 2.88 (1.56) | 3.62 (1.53) | 3.99 (1.38)
  Nausea and vomiting: Change at 12 months | 2.08 (1.34) | 2.05 (1.43) | 3.51 (1.26)
  Nausea and vomiting: Change at 24 months | 1.19 (1.19) | 0 (0) | 1.59 (1.09)
  Pain: Change at 3 months | 2.57 (4.03) | 1.63 (3.95) | 3.53 (3.56)
  Pain: Change at 12 months | 6.24 (3.89) | 4.41 (4.11) | 14.42 (3.64)
  Pain: Change at 24 months | 2.84 (4.84) | 2.12 (5.21) | 2.99 (3.92)
  Physical functioning: Change at 3 months | -1.68 (2.51) | -7.72 (2.46) | -3.87 (2.22)
  Physical functioning: Change at 12 months | -4.90 (2.45) | -6.32 (2.59) | -6.78 (2.30)
  Physical functioning: Change at 24 months | -7.08 (2.96) | -3.61 (3.21) | -3.80 (2.50)
  Role functioning: Change at 3 months | -6.92 (3.94) | -4.70 (3.87) | -8.14 (3.48)
  Role functioning: Change at 12 months | -6.55 (4.00) | -9.65 (4.24) | -12.12 (3.75)
  Role functioning: Change at 24 months | -3.48 (4.99) | 0.08 (5.43) | -7.57 (4.06)
  Social functioning: Change at 3 months | -5.72 (4.03) | -1.95 (3.96) | -9.57 (3.56)
  Social functioning: Change at 12 months | -6.95 (3.69) | -0.37 (3.91) | -5.01 (3.45)
  Social functioning: Change at 24 months | 5.15 (4.64) | 3.90 (5.06) | -2.93 (3.81)

4. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaire-Prostate 25 (QLQ-PR25) Score at 3, 12 and 24 Months
Description: EORTC QLQ-PR25, a module of the EORTC QLQ-30 questionnaire was used to assess the quality of life. It Consist of 25 questions distributed on 6 domains: urinary symptoms (8 items), incontinence aid (1 item), bowel symptoms (4 items), hormonal treatment-related symptoms (HTRS) (6 items), sexual activity (2 items), and sexual functioning (4 items). Participants answered each of these questions on a 4 point scale (1 'Not at all' to 4 'Very much'). All raw domain scores are linearly transformed to a 0-100 scale, with higher scores reflecting either more symptoms (urinary, bowel, hormonal treatment-related symptoms) or higher levels of activity or functioning (sexual).
Time Frame: Baseline, at 3, 12 and 24 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 30 | 29 | 31
Units on a scale
  Incontinence aid: Change at 3 months | 21.74 (11.72) | 3.35 (14.22) | 12.09 (10.97)
  Incontinence aid: Change at 12 months | 14.31 (9.92) | 15.11 (10.07) | 2.78 (9.44)
  Incontinence aid: Change at 24 months | 20.60 (16.04) | 32.59 (12.52) | 19.46 (9.82)
  Bowel symptoms: Change at 3 months | 1.43 (1.53) | 4.27 (1.49) | 5.37 (1.33)
  Bowel symptoms: Change at 12 months | 5.11 (1.57) | 1.36 (1.69) | 3.76 (1.45)
  Bowel symptoms: Change at 24 months | -0.82 (1.98) | 0.93 (2.09) | 1.48 (1.56)
  HTRS: Change at 3 months | 10.56 (2.25) | 8.09 (2.21) | 13.32 (2.01)
  HTRS: Change at 12 months | 14.72 (2.44) | 18.05 (2.59) | 19.43 (2.30)
  HTRS: Change at 24 months | 6.42 (3.16) | 1.30 (3.45) | 5.39 (2.62)
  Sexual activity: Change at 3 months | 20.18 (4.40) | 16.10 (4.32) | 19.78 (3.98)
  Sexual activity: Change at 12 months | 33.50 (4.03) | 19.16 (4.24) | 25.02 (3.83)
  Sexual activity: Change at 24 months | 13.17 (5.23) | 11.46 (5.72) | 12.56 (4.39)
  Sexual functioning: Change at 3 months | 9.65 (9.80) | 22.03 (9.03) | 37.20 (10.73)
  Sexual functioning: Change at 12 months | 10.65 (10.09) | -1.19 (9.05) | 10.73 (11.14)
  Sexual functioning: Change at 24 months | -6.41 (12.58) | 12.33 (11.54) | 0.32 (11.34)
  Urinary symptoms: Change at 3 months | 8.87 (2.61) | 2.55 (2.54) | 7.16 (2.28)
  Urinary symptoms: Change at 12 months | 5.47 (2.45) | 1.81 (2.57) | 10.54 (2.26)
  Urinary symptoms: Change at 24 months | 5.87 (3.26) | 0.52 (3.50) | 9.16 (2.70)

5. Secondary Outcome: Change From Baseline in Sexual Health Inventory for Men (SHIM) Total Score at 3, 12, 24 Months
Description: The SHIM is a well validated abridged 5-item of the 15-item International Index of Erectile Function, which has been extensively studied in men with erectile dysfunction due to various etiologies, including prostate cancer-related therapies. It consists of 5 items pertaining to sexual functioning, with scores ranging from 0-5 for most items. The total score is obtained by adding all five item scores, and can range from 5 to 25. Higher scores indicate higher level of sexual function and less erectile dysfunction.
Time Frame: Baseline, at 3, 12, 24 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 30 | 29 | 31
Units on a scale
  Change at 3 months | -3.64 (0.74) | -1.80 (0.67) | -3.54 (0.63)
  Change at 12 months | -3.52 (0.81) | -2.91 (0.83) | -3.79 (0.78)
  Change at 24 months | -1.97 (1.16) | -2.03 (1.17) | -2.39 (0.99)

6. Secondary Outcome: Time to Prostate Specific Antigen (PSA) Progression Based on Modified Prostate Cancer Clinical Trials Working Group (PCWG2) Criteria
Description: PSA progression was defined as a rise to greater than 50 percent (%) of the baseline serum PSA or rise of 2 nanogram per milliliter (ng/mL) or more above the nadir, whichever is higher, confirmed by repeat measurement at least 2 weeks later.
Time Frame: Up to 24 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 30 | 29 | 31
Months | 30.88 [22.54 to NA] — Here, NA indicates upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of events. | 25.79 [20.04 to 38.90] | 36.11 [26.97 to 56.64]

7. Secondary Outcome: Percentage of Participants Without PSA or Radiographic Progression and With Recovery of Serum Testosterone
Description: Percentage of participants without evidence of PSA or radiographic progression during the 24-month treatment period and with recovery of serum testosterone at 24 months were reported. Testosterone recovery was defined as a serum testosterone greater than (>) 150 nanogram per deciliter (ng/dL). PSA progression was defined as a rise to greater than 50 percent (%) of the baseline serum PSA or rise of 2 nanogram per milliliter (ng/mL) or more above the nadir, whichever is higher, confirmed by repeat measurement at least 2 weeks later. Radiographic progression was defined as the detection of new metastasis on either bone scan or cross-sectional imaging (computed tomography [CT] or magnetic resonance imaging [MRI]).
Time Frame: Up to 24 months
Population: Modified Intent-to-treat Population (mITT) included subset of ITT population for outcomes related to testosterone recovery, participants who withdrew from the study prior to 24 months after Day 1 were excluded from the analysis. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 26 | 27 | 29
Percentage of participants | 19.2 | 37.0 | 37.9

8. Secondary Outcome: Percentage of Participants With a Serum PSA Less Than 0.2 ng/mL
Description: Percentage of participants with PSA less than (<) 0.2 ng/mL after 7 months of protocol therapy were reported.
Time Frame: From 7 to 24 months
Population: mITT included subset of ITT population for outcomes related to testosterone recovery, participants who withdrew from the study prior to 24 months after Day 1 were excluded from the analysis. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 26 | 27 | 29
Percentage of participants | 88.5 | 88.9 | 96.6

9. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change from baseline in BMI was reported. BMI was calculated as 'body weight in kg/(height in meters)* (height in meters)'. Endpoint values are from the last measurement within the analysis period.
Time Frame: Baseline, Day 1 (Cycle 1), Day 28 (Cycle 1, 2, 4, 5, 7, 8, 10 and 11), Day 35 (Cycle 3, 6, 9 and 12) and endpoint (up to 24 months)
Population: The safety population included all participants who received at least 1 dose of study drug as actually treated. Here, 'n' (number of participants analyzed) signifies the number of participants analyzed at a specified time point. "Number Analyzed=0" signifies that no participants were evaluated for the specified parameter at that time point.
Measure: Mean (Standard Deviation); unit: Kilogram per meter square (kg/m^2)
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 29 | 29 | 31
Kilogram per meter square (kg/m^2)
  Change at Cycle 1 Day 1: number analyzed (Participants) | 1 | 0 | 1
  Change at Cycle 1 Day 1 | 0.00 |  | 0.00
  Change at Cycle 1 Day 28: number analyzed (Participants) | 27 | 27 | 31
  Change at Cycle 1 Day 28 | 0.00 (0.443) | -0.02 (0.569) | -0.29 (0.458)
  Change at Cycle 2 Day 28: number analyzed (Participants) | 28 | 27 | 31
  Change at Cycle 2 Day 28 | -0.06 (0.903) | -0.23 (0.616) | -0.32 (0.524)
  Change at Cycle 3 Day 35: number analyzed (Participants) | 28 | 26 | 31
  Change at Cycle 3 Day 35 | 0.02 (0.837) | -0.34 (0.729) | -0.24 (0.610)
  Change at Cycle 4 Day 28: number analyzed (Participants) | 27 | 28 | 31
  Change at Cycle 4 Day 28 | 0.19 (0.784) | -0.17 (0.710) | -0.12 (0.645)
  Change at Cycle 5 Day 28: number analyzed (Participants) | 26 | 28 | 30
  Change at Cycle 5 Day 28 | 0.26 (0.892) | -0.15 (0.830) | 0.05 (0.716)
  Change at Cycle 6 Day 35: number analyzed (Participants) | 26 | 26 | 30
  Change at Cycle 6 Day 35 | 0.43 (0.851) | -0.15 (1.041) | -0.01 (0.771)
  Change at Cycle 7 Day 28: number analyzed (Participants) | 25 | 26 | 29
  Change at Cycle 7 Day 28 | 0.48 (0.862) | -0.16 (1.114) | 0.07 (0.743)
  Change at Cycle 8 Day 28: number analyzed (Participants) | 25 | 26 | 30
  Change at Cycle 8 Day 28 | 0.56 (0.880) | 0.02 (1.208) | 0.15 (0.811)
  Change at Cycle 9 Day 35: number analyzed (Participants) | 25 | 26 | 30
  Change at Cycle 9 Day 35 | 0.58 (0.919) | 0.04 (1.189) | 0.06 (0.822)
  Change at Cycle 10 Day 28: number analyzed (Participants) | 24 | 26 | 30
  Change at Cycle 10 Day 28 | 0.66 (1.059) | 0.12 (1.345) | 0.20 (0.584)
  Change at Cycle 11 Day 28: number analyzed (Participants) | 25 | 26 | 29
  Change at Cycle 11 Day 28 | 0.63 (1.227) | 0.04 (1.248) | 0.24 (0.825)
  Change at Cycle 12 Day 35: number analyzed (Participants) | 25 | 25 | 29
  Change at Cycle 12 Day 35 | 0.66 (1.049) | 0.01 (1.312) | 0.15 (0.682)
  Endpoint: number analyzed (Participants) | 28 | 28 | 31
  Endpoint | 0.65 (0.992) | -0.07 (1.272) | 0.11 (0.705)

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: The change from baseline in fasting plasma glucose levels was analyzed and reported using a mixed-model for repeated measures.
Time Frame: Baseline, Day 35 (Cycle 3, 6, 9 and 12)
Population: The ITT population included all randomized participants and was classified according to their assigned treatment group, regardless of the actual treatment received. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Millimoles per liter (mmol/L)
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 29 | 29 | 31
Millimoles per liter (mmol/L)
  Change at Cycle 3 Day 35 | -0.07 (0.24) | 0.11 (0.23) | 0.61 (0.21)
  Change at Cycle 6 Day 35 | 0.19 (0.19) | -0.00 (0.19) | 0.27 (0.17)
  Change at Cycle 9 Day 35 | 0.10 (0.18) | -0.10 (0.19) | 0.41 (0.16)
  Change at Cycle 12 Day 35 | 0.29 (0.19) | 0.15 (0.19) | 0.26 (0.16)

11. Secondary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1C)
Description: The change from baseline in HbA1C was analyzed and reported using a mixed-model for repeated measures.
Time Frame: Baseline, Day 35 (Cycle 3, 6, 9 and 12)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1C
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 29 | 29 | 31
Percentage of HbA1C
  Change at Cycle 3 Day 35 | 0.14 (0.06) | -0.07 (0.06) | 0.06 (0.06)
  Change at Cycle 6 Day 35 | 0.09 (0.06) | -0.10 (0.06) | 0.08 (0.06)
  Change at Cycle 9 Day 35 | 0.16 (0.06) | -0.13 (0.06) | 0.04 (0.06)
  Change at Cycle 12 Day 35 | 0.18 (0.06) | -0.09 (0.06) | 0.13 (0.06)

12. Secondary Outcome: Change From Baseline in Cholesterol, High-density Lipoprotein (HDL) Cholesterol, Low-density Lipoprotein (LDL) Cholesterol and Triglycerides
Description: Change from baseline in cholesterol, HDL cholesterol, LDL cholesterol and triglycerides were analyzed and reported using a mixed-model for repeated measures.
Time Frame: Baseline, Day 35 (Cycle 3, 6, 9 and 12)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 29 | 29 | 31
mmol/L
  Cholesterol: Change at Cycle 3 Day 35 | 0.34 (0.16) | 0.98 (0.16) | 1.28 (0.13)
  Cholesterol: Change at Cycle 6 Day 35 | 0.18 (0.16) | 0.71 (0.16) | 1.35 (0.13)
  Cholesterol: Change at Cycle 9 Day 35 | 0.24 (0.16) | 0.66 (0.17) | 1.21 (0.14)
  Cholesterol: Change at Cycle 12 Day 35 | 0.38 (0.16) | 0.71 (0.17) | 0.92 (0.15)
  LDL Cholesterol: Change at Cycle 3 Day 35 | 0.08 (0.15) | 0.67 (0.15) | 0.91 (0.13)
  LDL Cholesterol: Change at Cycle 6 Day 35 | -0.03 (0.15) | 0.36 (0.15) | 0.87 (0.13)
  LDL Cholesterol: Change at Cycle 9 Day 35 | 0.01 (0.14) | 0.28 (0.15) | 0.69 (0.13)
  LDL Cholesterol: Change at Cycle 12 Day 35 | 0.07 (0.15) | 0.31 (0.16) | 0.57 (0.13)
  HDL Cholesterol: Change at Cycle 3 Day 35 | 0.08 (0.04) | 0.07 (0.05) | 0.13 (0.04)
  HDL Cholesterol: Change at Cycle 6 Day 35 | 0.09 (0.04) | 0.16 (0.05) | 0.12 (0.04)
  HDL Cholesterol: Change at Cycle 9 Day 35 | 0.10 (0.05) | 0.21 (0.05) | 0.17 (0.04)
  HDL Cholesterol: Change at Cycle 12 Day 35 | 0.12 (0.05) | 0.21 (0.06) | 0.12 (0.05)
  Triglycerides: Change at Cycle 3 Day 35 | 0.27 (0.14) | 0.31 (0.14) | 0.34 (0.12)
  Triglycerides: Change at Cycle 6 Day 35 | 0.21 (0.15) | 0.14 (0.15) | 0.52 (0.13)
  Triglycerides: Change at Cycle 9 Day 35 | 0.30 (0.15) | -0.01 (0.16) | 0.53 (0.14)
  Triglycerides: Change at Cycle 12 Day 35 | 0.43 (0.15) | 0.08 (0.16) | 0.28 (0.13)

13. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD)
Description: Change from baseline in BMD was assessed for femoral neck and lumber spine with DEXA scans.
Time Frame: Baseline, Cycle 12 Day 35
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Gram per centimeter square (g/cm^2)
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 29 | 29 | 31
Gram per centimeter square (g/cm^2)
  Femoral Neck | 0.00 (0.03) | 0.07 (0.03) | -0.02 (0.02)
  Lumbar Spine | 0.00 (0.02) | 0.01 (0.02) | -0.06 (0.02)

14. Secondary Outcome: Median Time to Serum Testosterone Recovery to Greater Than (>) 50 ng/dL (Non-castrate) and > 150 ng/dL
Description: The time to serum testosterone recovery to > 50 ng/dL and > 150 ng/dL from Month 13 to Month 24 of protocol therapy was reported.
Time Frame: Month 13 to Month 24
Population: mITT included subset of ITT population for outcomes related to testosterone recovery, participants who withdrew from the study prior to 24 months after Day 1 were excluded from the analysis. This outcome measure was planned to be analyzed and reported for LHRHa-based treatment arms.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | LHRHa + Apalutamide
Number analyzed (Participants) | 27 | 30
Months
  > 50 ng/dL | 18.89 [18.04 to 23.95] | 18.10 [17.91 to 24.05]
  > 150 ng/dL | 23.33 [18.14 to 24.87] | 23.98 [18.00 to 24.08]

15. Secondary Outcome: Change From Baseline in Serum Dihydrotestosterone (DHT) Levels
Description: Change from baseline in serum DHT levels was reported.
Time Frame: Baseline, Day 35 (Cycle 6 and Cycle 12)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Nanomoles per liter (nmol/L)
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 29 | 29 | 31
Nanomoles per liter (nmol/L)
  Change at Cycle 6 Day 35 | -0.90 (0.26) | 0.93 (0.27) | -0.90 (0.23)
  Change at Cycle 12 Day 35 | -0.90 (0.24) | 0.86 (0.25) | -0.90 (0.21)

16. Secondary Outcome: Change From Baseline in Estradiol Levels
Description: Change from baseline in estradiol levels was reported.
Time Frame: Baseline, Day 35 (Cycle 6 and Cycle 12)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Picomoles per liter (pmol/L)
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 29 | 29 | 31
Picomoles per liter (pmol/L)
  Change at Cycle 6 Day 35 | -88.63 (12.24) | 87.87 (13.37) | -94.11 (11.58)
  Change at Cycle 12 Day 35 | -77.12 (13.46) | 81.29 (13.88) | -103.01 (12.76)

17. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product. Treatment-emergent adverse events are those that occurred between the date of 1st dose of study drug and date of last dose of study drug plus 30 days.
Time Frame: From date of 1st dose of study drug to date of last dose of study drug plus 30 days (up to 6 years)
Population: The safety population included all participants who received at least 1 dose of study drug as actually treated.
Measure: Number; unit: Percentage of participants
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
Number analyzed (Participants) | 29 | 29 | 31
Percentage of participants | 96.6 | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Up to 6 years
Description: The safety population included all participants who received at least 1 dose of study drug as actually treated.
Arm/Group | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) | Apalutamide | LHRHa + Apalutamide
All-Cause Mortality (participants affected / at risk) | 1/29 | 0/29 | 0/31
Serious Adverse Events (participants affected / at risk) | 3/29 | 0/29 | 5/31
Other Adverse Events (participants affected / at risk) | 28/29 | 29/29 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) (N=29) | Apalutamide (N=29) | LHRHa + Apalutamide (N=31)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1
Device Failure (Product Issues) | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Toxic Epidermal Necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Luteinizing Hormone Releasing Hormone Agonist (LHRHa) (N=29) | Apalutamide (N=29) | LHRHa + Apalutamide (N=31)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 3 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 2
Eyelid Ptosis (Eye disorders) | 0 | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 5 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 3 | 4
Constipation (Gastrointestinal disorders) | 2 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 7 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 2
Flatulence (Gastrointestinal disorders) | 0 | 4 | 3
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 4 | 7
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3
Asthenia (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 22 | 19 | 24
Oedema Peripheral (General disorders) | 0 | 1 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 3 | 4
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 4
Aspartate Aminotransferase Increased (Investigations) | 2 | 0 | 0
Heart Rate Irregular (Investigations) | 0 | 2 | 0
Weight Decreased (Investigations) | 0 | 1 | 2
Weight Increased (Investigations) | 3 | 2 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 4 | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 8 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Cognitive Disorder (Nervous system disorders) | 0 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 4 | 4
Dysgeusia (Nervous system disorders) | 0 | 6 | 5
Headache (Nervous system disorders) | 0 | 2 | 6
Memory Impairment (Nervous system disorders) | 0 | 2 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 2 | 1
Depression (Psychiatric disorders) | 1 | 3 | 4
Insomnia (Psychiatric disorders) | 2 | 1 | 10
Irritability (Psychiatric disorders) | 2 | 0 | 0
Libido Decreased (Psychiatric disorders) | 3 | 1 | 3
Loss of Libido (Psychiatric disorders) | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 1 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 2
Breast Tenderness (Reproductive system and breast disorders) | 0 | 4 | 2
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 3 | 1
Gynaecomastia (Reproductive system and breast disorders) | 3 | 12 | 1
Nipple Pain (Reproductive system and breast disorders) | 0 | 12 | 0
Testicular Pain (Reproductive system and breast disorders) | 2 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 4 | 3
Hypotrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 5
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Hot Flush (Vascular disorders) | 25 | 9 | 26
Hypertension (Vascular disorders) | 0 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT01790126/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/26/NCT01790126/SAP_001.pdf